CLINICAL TRIAL: NCT05860478
Title: Wearable Technology for Promoting Physical Activity in Middle-Aged Adults With Chronic Musculoskeletal Pain
Brief Title: Wearable Device to Increase Physical Activity Amongst Adults With Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West London (Other)
Collaborators: Royal London Hospital for Integrated Medicine (Other)
Responsible Party: Principal Investigator, John Hughes, Associate Professor, University of West London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 314666
Record Dates: First submitted 2023-04-07; First posted 2023-05-16 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Musculoskeletal Chronic Pain Conditions
MeSH Terms: interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wearable device plus standard care (Experimental)
  Interventions: Device: Wearable device
- standard care (No Intervention)

INTERVENTIONS:
Device: Wearable device — The wearable device includes a motion sensor, and is worn around the wrist, and the device records a participant's physical activity .
  Arms: wearable device plus standard care

SUMMARY:
This protocol is for a pragmatic mixed methods randomized parallel-group exploratory feasibility trial to examine all facets of a proposed future phase III trial on the use of wearable device to increase physical activity and possibly reduce pain amongst middle-aged people with musculoskeletal (MSK) chronic pain. The feasibility study is intended to answer the following research questions:

Question 1 Evaluate the acceptability of all aspect of the study design of wearable devices as an intervention to increase physical activity in middle-aged adults with musculoskeletal chronic pain.

Question 2: Is it feasible and acceptable to use wearable devices as an intervention to increase physical activity in middle-aged adults with musculoskeletal chronic pain? Question 3: How can using wearable device promote physical activity effectively in middle-aged adults with musculoskeletal chronic pain?

Participants will be recruited from a National Health Service (NHS) pain clinic and randomised on a ratio1:3 into control group (standard care) and intervention group (standard care combined with wearable device). The feasibility study will last for 18 months, participants involvement will be for 24 weeks. Patients in both groups can participate in any physical activity, including planned, structured, and repetitive bodily movement exercise or occupational and recreational PA. Qualitative semi-structured interview will be conducted at baseline and week-12, while outcome measures will be conducted at baseline, 4-week, 8-week,12-week, and 24-week for all participants to examine their pain, physical activity, and their responses to the trial. Qualitative interview will be conducted for stakeholders which include clinicians and service managers after all patient data has been collected. This study has the potential to make an original contribution to provide key data on the feasibility, acceptability, and effectiveness of using wearable technology to support physical activity intervention for middle-aged adults with musculoskeletal chromic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient of any gender identity 40-65 years old.
* Willingness to participate in the trial.
* Able to understand and speak sufficient English to engage during interviews.
* They have self-reported persistent or recurrent musculoskeletal pain for three months or longer.
* Participants will be receiving treatment for musculoskeletal chronic pain.

Exclusion Criteria:

* Palliative patient.
* Patients of any gender identity younger than 40-year-old or older than 65-year-old.
* Patients that are dependent on alcohol or drugs.
* Involvement with other ongoing studies.
* Patients unable to complete the questionnaires as judged by the researcher.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Pain Inventory | Participants in both groups will complete outcome measures at baseline (T0), week 4 (T1), week 8 (T2), week 12 (T3), and week 24 (T4)
Change in Visual Analogue Scale (VAS) of Quality of Life | Participants in both groups will complete outcome measures at baseline (T0), week 4 (T1), week 8 (T2), week 12 (T3), and week 24 (T4)
Change in Visual Analogue Scale (VAS) of pain | Participants in both groups will complete outcome measures at baseline (T0), week 4 (T1), week 8 (T2), week 12 (T3), and week 24 (T4)
Change in Numerical Pain Rating Scale (NPRS) | Participants in both groups will complete outcome measures at baseline (T0), week 4 (T1), week 8 (T2), week 12 (T3), and week 24 (T4)
Change in EuroQol Five-Dimensional Questionnaire (EQ-5D-5L) | Participants in both groups will complete outcome measures at baseline (T0), week 4 (T1), week 8 (T2), week 12 (T3), and week 24 (T4)
Change in Pain Catastrophising Scale | Participants in both groups will complete outcome measures at baseline (T0), week 4 (T1), week 8 (T2), week 12 (T3), and week 24 (T4)
Change in The International Physical Activity Questionnaire (IPAQ) | Participants in both groups will complete outcome measures at baseline (T0), week 4 (T1), week 8 (T2), week 12 (T3), and week 24 (T4)
Change in Chronic Pain Coping Inventory (CPCI) | Participants in both groups will complete outcome measures at baseline (T0), week 4 (T1), week 8 (T2), week 12 (T3), and week 24 (T4)
Change in Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) | Participants in both groups will complete outcome measures at baseline (T0), week 4 (T1), week 8 (T2), week 12 (T3), and week 24 (T4)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital for Integrated Medicine, UCLH NHS Foundation Trust, London, United Kingdom